CLINICAL TRIAL: NCT00449592
Title: A Ramdomized Double Blined Placebo Controlled Oral Zinc Therapy for the Prevention of Mucositis in Patients Undergoing High Dose Chemotherapy With Stem Cell Support
Brief Title: Oral Zinc Therapy for the Prevention of Mucositis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Maya Koren-Michovitz, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SHEBA-06-4196-MKM-CTIL
Record Dates: First submitted 2007-03-18; First posted 2007-03-20 (Estimated); Last update posted 2008-10-03 (Estimated); Status verified 2008-10

CONDITIONS: Mucositis
Keywords: Stem cell transplantation; Mucositis; Zinc
MeSH Terms: conditions — Mucositis | interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Oral zinc therapy, intervention
  Interventions: Drug: Zinc
- 2 (Placebo Comparator): oral placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zinc — Oral Zincol 1 Tab TID from day -6/-7 until discharge
  Arms: 1
Drug: Placebo — Oral placebo 1 Tab TID from day -6/-7 until discharge
  Arms: 2

SUMMARY:
Zinc is an intracellular mineral with important enzymatic cofactor activities for cell membrane stability, DNA and RNA structure. Zinc deficiency is associated with delayed wound healing and immune dysfunction. In patietns with hematological malignancies an inverse correlation was found between disease stage and zinc level. Patients undergoing high dose chemotherapy for hematologic malignancies are predisposed to develop oral and gastrointestinal complications, in particular oral mucositis. These patients may have relative zinc deficiency, therefore oral zinc therapy may be benefical in the prevention of these complications.

DETAILED DESCRIPTION:
Patients candidate for High dose chemotherapy with stem cell support for the diagnosis of relapsed/resistant Hodgkins or NHL or MM will be screened for enrollment in the study.

Patients will be randomized in a 1:1 ratio to therapy with either zincol 1 Tab TID or placebo 1 Tab TID.

Therapy will start on the morning before commencing chemotherapy and will continue untill the first of either discharge day or day 21.

Response assesment will include:

1. Mucositis assesment using NCI-CTC and OMAS scores- to be done eod from baseline and untill day 21/discharge day if before day 21
2. Evaluation of zinc levels in the serum, PBMC and saliva- to be done at baseline, day 6/7 and day 21/discharge day if before day 21.
3. Collection of clinical outcome data regarding infectious complications including- presence and length of febrile neutropenia,use of antibacterial and antifungal medications,

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing high dose chemotherapy with stem cell support for relapsed or resistant Hodgkins or NHL (treated with BEAM protocol) or MM (treated with high dose melphalan).
* ECOG performance less than or equal to 2
* Adequate renal and hepatic function

Exclusion Criteria:

* Presence of any other active malignancy other than BCC of the skin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Maximal Mucositis grade | day -7 to day +21 or discharge day

SECONDARY OUTCOMES:
Duration of maximal mucositis grade | day -7 to day +21 or discharge day
Overall duration of mucositis | day -7 to day +21 or discharge day
Duration of severe neutropenia | day -7 to day +21 or discharge day
Duration of febrile neutropenia | day -7 to day +21 or discharge day

CONTACTS AND LOCATIONS:
Overall Officials: Maya Koren-Michowitz, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Division of Hematology and Bone Marrow Transplantation, Sheba Medical Center, Ramat Gan, Israel